CLINICAL TRIAL: NCT01436942
Title: Effect of Exercise on Disease Activity and Cardiovascular Risk Factors in Patients With AS: A Single Blind Randomized Controlled Trail
Brief Title: Effect of Exercise on Disease Activity and Cardiovascular Risk Factors in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Silje H Sveaas, PT, PhD, PhD.student, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Diakonhjemmet Hospital
Record Dates: First submitted 2011-09-13; First posted 2011-09-20 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2013-03

CONDITIONS: Ankylosing Spondyliti
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Experimental)
  Interventions: Behavioral: Exercise
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — The exercise intervention will be carried out at a fitness center with supervision from a physiotherapist.
  A cardiorespiratory and muscle strengthening exercise program following the American College of Sports Medicine (ACSM) recommendations for maintenance and improvement of physical fitness. Cardiorespiratory fitness: two interval sessions (4 x 4 min), one continuous moderate exercise session (40 min) on a treadmill. The muscle strength exercises will consist of: 15-20 repetitions, large muscle groups as thighs, back and abdomen.
  Dose: 12 weeks. Three times a week, 60 minutes.
  Arms: Exercise group

SUMMARY:
Background:

Exercise is recommended as a cornerstone in the treatment of ankylosing spondylitis together with medication. Last years, increased risk of cardiovascular diseases in patient with inflammatory diseases is reported, probably caused by inflammation and increased prevalence of traditional risk factors. In both healthy adults and other patient groups, cardiorespiratory and muscular strength exercises have been shown to have a positive effect on inflammation as well as on cardiovascular risk factors. To our knowledge this has not been shown in patients with ankylosing spondylitis.

Objective: The aim of this study is to investigate the effects of a cardiorespiratory and muscular strength exercise program on disease activity and cardiovascular risk factors in patients with ankylosing spondylitis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis, confirmed by a rheumatologist
* Age, 18-70 years
* Not using TNF-α medication or steady medication for ≥3 months
* Disease activity ≥2.1 on ankylosing spondylitis disease activity score defined as high disease activity
* Not participated in a structured cardiorespiratory or muscle strengthening exercise program during the last year (>60 min once per week), including large amounts of brisk walking (>120 min per week)

Exclusion Criteria:

* Known cardiovascular disease
* Severe comorbidity which involves reduced exercise capacity
* Not able to participate in weekly exercises sessions in Oslo
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Disease activity | 12 weeks after baseline assessment
  The Ankylosing Spondylitis Disease Activity Score-C-reactive protein (ASDAS-CRP) will be used to assess disease activity. It is a continuous measure based on patient-reported outcomes (back pain, duration of morning stiffness, patient global assessment and peripheral join complaints) and CRP, and higher values indicate higher disease activity. The minimal clinically important improvement for this instrument is reported to be ∆ ≥1.1, and ∆ ≥2.0 is considered a major improvement.

SECONDARY OUTCOMES:
Electrocardiography | 12 weeks after baseline assessment
  To measure the electrical activity of the heart.
Blood samples | 12 weeks after baseline assessment
  Analyzed for both general and endothelial specific markers of inflammation and cardiovascular risk(total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, glucose, NTproBNP, TNF-α, IL-6, IL-18, high sensitive C-reactive protein and sedimentation rate)
Blood pressure | 12 weeks after baseline assessment
Physical fitness | 12 weeks after baseline assessment
  Cardiorespiratory fitness will be assessed with an indirect maximal walking test on a treadmill for estimation of peak oxygen uptake according to modified Balke protocol. Hand grip strength will be assessed with GRIPPIT. Spinal and hip mobility will be assessed with the Bath Ankylosing Spondylitis Metrology index (BASMI), and chest expansion will be measured as the difference between maximal inspiration and expiration at the level of xipoideus (cm).
Body composition | 12 weeks after baseline assessment
  Weight, height, waist circumference will be measured. Dual Energy X-ray Absortiometry (DEXA) will be used to assess body composition.
Physical function | 12 weeks after baseline assessment
  Will be assessed with the patient reported index Bath Ankylosing Spondylitis Functional Index (BASFI).
General health | 12 weeks after baseline assessment
  Will be assessed with the generic General Health Questionnaire (GHQ-12).
Physical activity level | 12 weeks after baseline assessment and 12 months after the intervention
  Will be assessed with the International Physical Activity Questionnaire short version (IPAQ-s).

CONTACTS AND LOCATIONS:
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

REFERENCES:
- [Derived] Sveaas SH, Berg IJ, Provan SA, Semb AG, Hagen KB, Vollestad N, Fongen C, Olsen IC, Michelsen A, Ueland T, Aukrust P, Kvien TK, Dagfinrud H. Efficacy of high intensity exercise on disease activity and cardiovascular risk in active axial spondyloarthritis: a randomized controlled pilot study. PLoS One. 2014 Sep 30;9(9):e108688. doi: 10.1371/journal.pone.0108688. eCollection 2014. PMID 25268365